CLINICAL TRIAL: NCT06100679
Title: Responsible Engaged and Loving (REAL) Fathers: Study Protocol for a Cluster-randomized Controlled Trial of Mentored Parenting Sessions for Young Fathers to Promote Child Development and Reduce Violence in Uganda
Brief Title: Responsible Engaged and Loving (REAL) Fathers Intervention Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Impact and Innovations Development Centre (IIDC), Uganda (Unknown); NaNa Development Consultants Ltd, Uganda (Unknown); LEGO Foundation (Unknown)
Responsible Party: Principal Investigator, Kathryn Barker, Assistant Professor, Division of Infectious Diseases and Global Public Health, University of California, San Diego
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 808321
Record Dates: First submitted 2023-10-06; First posted 2023-10-25 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Violence, Gender-Based; Violence, Domestic; Violence, Sexual; Violence, Physical; Contraception Behavior; Child Development; Child Abuse; Communication, Partner; Conflict Resolution; Parent-Child Relations
Keywords: Violence Prevention; Early Childhood Development; Couples Communication; Father Engagement; Gender Norms
MeSH Terms: conditions — Coitus; Contraception Behavior; Communication; Negotiating

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized controlled trial-sequential transition of clusters from control to intervention conditions in randomized order, until all clusters are exposed.
Who Masked: Outcomes Assessor
Masking Description: Trained enumerators will be blinded to the treatment conditions from the beginning of the study (i.e., at baseline data collection) and before entering clusters (i.e., villages/communities) at mid-term and endline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care. Participants will have access to existing health centers and early childhood development centers.
- Intervention (Experimental): Participants will engage in the Responsible, Engaged and Loving (REAL) Fathers Intervention-an evidence-based community mentoring education program for young fathers and their spouses. Over 7 months, fathers receive monthly home visits from a community-identified male mentor. Mentors share information and skills-building tools on conflict resolution, non-violent discipline, family planning, and couple communication. At the end of each month, pairs or trios of mentors hold group reflection sessions with all mentored fathers. In months 5 and 6 of the intervention, spouses join the home visits and group sessions. Community-level intervention components include: 1) monthly educational poster campaigns that showcase nonviolent discipline and conflict resolution strategies; 2) community-hosted celebrations at the end of the intervention to acknowledge the accomplishments of the young fathers.
  Interventions: Behavioral: Responsible Engaged and Loving (REAL) Fathers Initiative

INTERVENTIONS:
Behavioral: Responsible Engaged and Loving (REAL) Fathers Initiative — REAL Fathers is a multilevel norms-shifting intervention among: young fathers (ages 16-25 whose oldest child is under the age of 3); couple dyads (fathers and wives); mentoring dyads and groups; and communities. Respected men in the community are identified by participating young fathers, their partners and community members to become mentors. Mentors participate in a training and mentor young fathers through home and group sessions on conflict resolution, non-violent discipline, family planning, and couple communication. Mentoring is supplemented with a monthly poster campaign designed to reinforce messages from the home and group mentoring sessions and a community celebration. REAL Fathers aims to build positive partnerships and parenting practices among young fathers to: 1) reduce incidence of intimate partner violence; 2) reduce harsh physical punishment of children; 3) improve early childhood development; 4) decrease unmet need for family planning.
  Other Names: REAL Fathers
  Arms: Intervention

SUMMARY:
The goal of this stepped-wedge cluster randomized control trial is to assess whether a Ugandan community-based intervention for young fathers (ages 18-25 years) of children ages 0-3 years impacts fathers' knowledge, attitudes, and behaviors surrounding positive parenting practices, father-child interaction, harsh physical punishment of children, and intimate partner violence.

DETAILED DESCRIPTION:
1. BACKGROUND. The prevalence of violence against women and children in Uganda takes a substantial toll on the overall health and welfare of families. Globally three in four children aged 2 to 4 years are exposed to harsh physical punishment. Child maltreatment not only inflicts immediate harm but also has long-lasting consequences on a child's physical and mental health, educational attainment, and overall development. One in four children under the age of five live with a mother who is a victim of intimate partner violence. Based on data from recent population surveys, 60% of Ugandan women reported having experienced intimate partner violence (IPV) at some point, while 45% reported experiencing IPV within the past year. These statistics underscore the urgent need for effective measures to address and mitigate the impact of such violence on the well-being of individuals and families in Uganda.
2. INTERVENTION. The Responsible, Engaged and Loving (REAL) Fathers Initiative is an evidence-based father-centered mentoring program designed to address social and gender norms that promote use of violence in child discipline and with intimate partners through promotion of positive parenting and partnership skills building. The REAL Fathers Initiative uses a 7-month mentoring program and a community poster campaign to model alternative strategies for nonviolent discipline and conflict resolution to improve fathers' parenting and communication skills and confidence in adapting nonviolent strategies. The project works with young fathers (ages 18-25) who have toddler-aged children (0-3 years) who are learning new roles as parents and husbands. This stage in a man's life is an ideal time to promote nonviolence in parenting and partner relationships as there is still ambiguity in the normative expectations about these roles and behaviors.
3. STUDY DESCRIPTION. This study will examine the impacts of a multilevel community-based intervention for young fathers and their families in Uganda on positive parenting, childhood development, and violence reduction. We will use a stepped-wedge cluster-randomized controlled trial design within 72 sub-counties randomly sampled from 24 districts in six regions of Uganda. Sub-counties are randomly allocated to treatment or control conditions at three successive time points from November 2023 to December 2025. Study participants are couple dyads (young fathers and their wives) ages 16-25 years with children ≤3 years (n=3,744 dyads). Quantitative longitudinal data will be collected via trained enumerators in six local languages on KoboCollect software. Intervention effects on primary and secondary outcomes will be assessed using difference-in-differences statistical approaches in mixed-effects models that account for the clustered stepped-wedge design.

ELIGIBILITY:
Inclusion Criteria for Young Fathers:

* Living in one of the six selected regions and districts across each region
* Being male aged between aged 16-25 years
* Being biological father to a child(ren) who is younger than 3 years old
* Living in union and in the same household with the mother or guardian of the child(ren)

Inclusion Criteria for Spouses:

* Living in union and in the same household as the young father

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4728 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Reduced Intimate Partner Violence Perpetration (IPV-P) | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of young fathers and their wives reporting perpetrating physical, sexual, and/or emotional IPV in the past three months. Assessed via six measures: whether you shouted or yelled at your [wife/husband]; slapped your [wife/husband]; pushed or shoved your [wife/husband]; threw something at your [wife/husband] that could hurt [her/him]; physically forced your [wife/husband] to have sex with you when [she/he] did not want to; or insulted your [wife/husband]. Response options: never, once, a few times, many times, don't know/remember, refused.
Reduced Intimate Partner Violence Victimization (IPV-V) | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of young fathers and their wives reporting being a victim of physical, sexual, and/or emotional IPV in the past three months. Six measures include: whether your spouse shouted or yelled at you; slapped you; pushed or shoved you; threw something at you that could hurt you; physically forced you to have sex with you when you did not want to; or insulted you. Response options: never, once, a few times, many times, don't know/remember, refused.
Reduced Unmet Need for Family Planning | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of men and women with unmet need for healthy timing and spacing of children. Assessed via those who are fecund and sexually active but are not using any method of contraception, and report not wanting any more children or wanting to delay the next child for 2 or more years.
Early Child Development (ECD) - CREDI | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Scores on the short-form version of the Caregiver Reported Early Development Instruments (CREDI).
Father engagement in child immunization | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of fathers reporting that they took their child(ren) for rounds of immunization(s).

SECONDARY OUTCOMES:
Fathers' knowledge of positive parenting and discipline skills | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of fathers who can correctly distinguish between positive and harsh parenting/ discipline. Item: There are various ways parents can use to positively disciple their children. Please tell me which of the following are positive ways parents can discipline their children. a) Taking a deep breath (calming yourself) when the child does something wrong before responding; b) Threaten to hit him/her; c) Tell your wife to take care of the child; d) Put him/her somewhere by him/herself; e) Redirect child's attention or behavior; f) Asking your wife for her advice or help; g) Shouting at him/her. Response options: True, False, Don't know, Refused
Fathers' attitudes towards positive parenting and discipline | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of fathers who hold positive attitudes for the use of non-violent parenting practices. Questions include: Stubborn children need to be hit to teach them right from wrong [reverse-coded].; A parent should never spank or hit a child.; Being violent with my child(ren) is not the only way to be an effective head of the family.; If a child is old enough to defy a parent, then he/she is old enough to be hit. [reverse-coded] Response options: strongly agree, agree, neither agree nor disagree, disagree, strongly disagree, don't know, refused.
Father engagement at home | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of young fathers who engage with household chores and caretaking activities in past three months. Items include: washed clothes; prepared food; bought food; played with your children at home; cooked or fixed food for your child; dressed or changed the clothes of the child; gave your child a bath; read books or looked at the pictures in books with the child; told stories to the child; sang songs with the child; took the child outside the home, compound, yard, or enclosure; spent time with the child naming, counting, and/or drawing things. Response options: never, rarely, once or twice a month, several times a week, every day, don't know/remember, refused.
Couple communication and conflict resolution | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of young fathers reporting increased and improved communication with their wives. Questions include whether in the past month the young father: took time to listen to his wife's concerns; communicated with each other about things that frustrated you; talked about things that affect each other and the family; and asked questions and got feedback/input from each other before making final decisions; resolved conflicts/arguments amicably without physically hurting each other. Response options: yes, no, don't know, refused.
Fathers' positive parenting and discipline behaviors | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of fathers reporting use of positive parenting and discipline practices in the past three months. Questions include: whether the father said something nice about or praised the child; gave the child physical affection; went someplace or did something special with the child as a reward; showed or told the child that you love him/her. Discipline strategies include: taking away something the child liked; explaining why the child's behavior was wrong; redirecting (giving the child something else to do); asking the child to apologize. Response options include: never, once, a few times, many times, don't know/remember, refused.
Reduced harsh violent discipline of children | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of fathers reporting they used a form of harsh/violent discipline with their child in the past month. Items include: shook child; shouted, yelled at, or screamed at child; spanked, hit, or slapped child on the bottom with bare hand; hit child on the bottom or elsewhere on the body with something like a belt, stick, or other hard object; hit or slapped child on the face, head, or ear; hit or slapped child on the hand, arm, or leg; beat child up, that is, hit him/her over and over as hard as you could. Response options: never, once, a few times, many times, don't know/remember, refused.
Supportive environments for father engagement and positive parenting | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of fathers agreeing or strongly agreeing that their social networks approve of engaging with children and using positive parenting skills. Items include: Your closest friends will tease you if you help your wife with child care. [reverse-coded] ; Your father would admire you for telling stories to your child(ren).; You would be embarrassed if your mother saw your child(ren) misbehave and you did not discipline the child strongly. [reverse-coded]; Your friends think you should discipline your child(ren) with love.; Your respected community members will say you are not parenting your child well if - instead of beating your child - you try to explain to them their misbehavior. [reverse-coded] Response options: strongly agree, agree, neither agree nor disagree, disagree, strongly disagree, don't know, refused.
Knowledge of where to access family planning method(s) | 1) Baseline to Wave 2 (Endline) = 8 months; and 2) Baseline to Wave 3 (Follow-Up) = 16 months
  Proportion of fathers and their wives who know where to obtain a method of family planning.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Barker, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (4):
- Uganda (4):
  - All Nations, Lira, Dokolo
  - Forum for African Women Educationalists (FAWE) - Uganda Chapter, Mbarara, Isingiro
  - Somero Uganda, Kampala, Kayunga, Bugiri, Luweero
  - Bantwana Initiatives Uganda, Kampala, Masindi, Kiryandongo and Katakwi

IPD SHARING:
Plan to Share IPD: Yes
Due to the highly sensitive nature of the resulting data on violence against children and women, these data will be available only through request to the study PI, who will vet requests to be certain that appropriate IRB approvals and data safety guidelines are in place.
Supporting Information: Study Protocol, ICF
Time Frame: Baseline data will become available Summer 2024; Endline data will become available Summer 2026.
Access Criteria: Appropriate IRB approvals and data safety guidelines.

REFERENCES:
- [Derived] Barker KM, Wandiembe S, Wandega A, Jeong J, Ojamuge D, Lundgren R, Yiga D, Nabembezi D. Testing the effectiveness of the Responsible, Engaged, and Loving Fathers (REAL Fathers) intervention for improving early childhood development and reducing family violence in Uganda: Study protocol for a cluster-randomized controlled trial. Trials. 2025 Sep 29;26(1):372. doi: 10.1186/s13063-025-09061-9. PMID 41024259